CLINICAL TRIAL: NCT00665951
Title: The Pharmacokinetics of Two Generic Co-formulations of Lopinavir/Ritonavir for HIV Infected Children: a Pilot Study of Lopimune vs. the Branded Product (SURF Study).
Brief Title: Pharmacokinetic Study of Two Generic Co-formulations of Lopinavir/Ritonavir for HIV Infected Children (SURF)
Acronym: SURF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Dr. D.M. Burger, hospital pharmacist, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 07.04
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections
Keywords: pediatric; pharmacokinetics; HIV infection
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Kaletra tablets
  Interventions: Drug: Lopinavir/ritonavir
- B (Experimental): Lopimune granules
  Interventions: Drug: Lopinavir/ritonavir
- C (Experimental): Lopimune tablets
  Interventions: Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir — Lopinavir/ritonavir 200/50mg; 2 tablets; single dose
  Other Names: Kaletra
  Arms: A
Drug: Lopinavir/ritonavir — Lopinavir/ritonavir 100/25mg; 4 sachets with granules; single dose
  Other Names: Lopimune granules
  Arms: B
Drug: Lopinavir/ritonavir — Lopinavir/ritonavir 100/25mg; 4 tablets; single dose
  Other Names: Lopimune tablets
  Arms: C

SUMMARY:
This pilot pharmacokinetic study is designed to exclude a large difference (>40%) in pharmacokinetics (esp. AUC) between two new Lopimune formulations and the branded formulation. The formal bioequivalence study with adequate power will be conducted by the manufacturer. In order to get data independently from the manufacturer and to have this information in an earlier phase, this small pilot study is initiated.

The initial study showed a declined bioavailability of the granules under fasting conditions. The study has been extended with an arm determining the pharmacokinetics of the granules after food (compared to the oral solution taken with food).

DETAILED DESCRIPTION:
Cipla has developed two co-formulated forms of lopinavir/ritonavir for second-line antiretroviral therapy for children: Lopimune granules and Lopimune tablets. They contain 100mg lopinavir and 25mg ritonavir.

Primary objective of this study:

To determine the pharmacokinetic profile of lopinavir and ritonavir in two different co-formulations (Lopimune granules and Lopimune tablets) after single-dose in HIV-negative, healthy adult subjects, and to compare this to the branded product.

Secondary objective:

To evaluate the safety of single-dose administration of the two generic co-formulations of lopinavir/ritonavir and compare this to the branded product.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years of age on the day of the first dosing.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first dosing.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age appropriate health condition
* Subject has a normal blood pressure and pulse rate, according to the investigator's judgment.
* Female subject is either not of childbearing potential, or is of childbearing potential and practicing one of the following methods of birth control: condoms, sponge, foams, jellies, diaphragm or copper intrauterine device (IUD); has a vasectomized partner; or total abstinence from sexual intercourse.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Therapy with any drug, including oral contraceptives.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), gastrointestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose.
* Pregnancy or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of lopinavir and ritonavir. | 0 (predose), 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 24 and 32 hours post ingestion (11 samples) on Days 1, 8 and 15.

SECONDARY OUTCOMES:
safety: adverse events | entire study

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] de Kanter CT, Colbers EP, Fillekes Q, Hoitsma A, Burger DM. Pharmacokinetics of two generic co-formulations of lopinavir/ritonavir for HIV-infected children: a pilot study of paediatric Lopimune versus the branded product in healthy adult volunteers. J Antimicrob Chemother. 2010 Mar;65(3):538-42. doi: 10.1093/jac/dkp472. Epub 2010 Jan 7. PMID 20056686